CLINICAL TRIAL: NCT05878548
Title: Management of Combined Fracture Neck of Femur and Femoral Deformity in Osteogenesis Imperfecta Patient
Acronym: OI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hesham Mohamed Elbaseet, Dr., Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOFOI
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis imperfecta; fracture neck of femur; telescoping nail
MeSH Terms: conditions — Osteogenesis Imperfecta; Femoral Neck Fractures

STUDY DESIGN:
Intervention Model Description: fixation with Wagner technique
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fixation with Wagner technique and Telescoping nail (Experimental): corrective osteotomy and intramedullary telescoping nail for deformed femur and Wagner technique to fix NOF fracture
  Interventions: Procedure: corrective osteotomy and intramedullary telescoping nail for deformed femur and Wagner technique to fix NOF fracture

INTERVENTIONS:
Procedure: corrective osteotomy and intramedullary telescoping nail for deformed femur and Wagner technique to fix NOF fracture — corrective osteotomy and intramedullary telescoping nail for deformed femur and Wagner technique to fix NOF fracture

SUMMARY:
O.I with NOF fixed by Wagner technique and telescoping nail

DETAILED DESCRIPTION:
osteogenesis imperfecta (Sillence Type IV) sustained neck of femur fracture after fall on ground. He had proximal femoral anterolateral bowing on top of inserted rod 4 years ago. He was treated with corrective osteotomy and intramedullary telescoping nail for deformed femur and Wagner technique to fix NOF fracture. One year after operation the patient gained satisfactory functional outcome with union of NOF fracture and correction of femoral deformity. This rare case illustrates the anticipated difficulties in managing neck of femur fracture in osteogenesis imperfect patients. The method of fixation with Wagner technique can achieve stable fixation for solid healing in fragility fractures like this and the least interference with telescoping nail insertion.

ELIGIBILITY:
Inclusion Criteria:

* OI

Exclusion Criteria:

* Not receiving Bisphosphonate

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
modified McKay's criteria | 1 year
  hip function score the higher the score the better outcome graded into excellent, Good , Fair and Poor

CONTACTS AND LOCATIONS:
Overall Officials: Hesaham M Elbaseet, MD, Principal Investigator — Assiut University
Locations (1):
- faculty of medicine Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hidalgo Perea S, Green DW. Osteogenesis imperfecta: treatment and surgical management. Curr Opin Pediatr. 2021 Feb 1;33(1):74-78. doi: 10.1097/MOP.0000000000000968. PMID 33278111
- [Background] Fralinger DJ, Kraft DB, Rogers KJ, Thacker MM, Kruse RW, Franzone JM. The Fate of the Bent Rod in Children With Osteogenesis Imperfecta. J Pediatr Orthop. 2023 Jul 1;43(6):e465-e470. doi: 10.1097/BPO.0000000000002409. Epub 2023 Apr 6. PMID 37026790